CLINICAL TRIAL: NCT01212185
Title: Oxytocin Treatment of Alcohol Withdrawal
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Principal Investigator, Cort Pedersen, MD, Professor, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 09-0172
Record Dates: First submitted 2010-09-28; First posted 2010-09-30 (Estimated); Results first posted 2014-05-13 (Estimated); Last update posted 2014-05-13 (Estimated); Status verified 2014-04

CONDITIONS: Alcohol Withdrawal
Keywords: oxytocin; alcohol withdrawal; lorazepam; alcoholism; intranasal administration; CIWA-Ar
MeSH Terms: conditions — Alcoholism | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- intranasal spray without oxytocin (Placebo Comparator): Twice daily intranasal spray without oxytocin.
  Interventions: Other: intranasal spray without oxytocin
- intranasal oxytocin spray (Experimental): Twice daily intranasal oxytocin spray
  Interventions: Drug: intranasal oxytocin spray

INTERVENTIONS:
Drug: intranasal oxytocin spray — 6 insufflations (24 IU of oxytocin total) given twice daily for 3 days
  Other Names: Syntocinon Spray
  Arms: intranasal oxytocin spray
Other: intranasal spray without oxytocin — 6 insufflations (0.1 metered dose/insufflation) twice daily
  Arms: intranasal spray without oxytocin

SUMMARY:
Purpose: Test whether intranasal administration of the neuropeptide, oxytocin, is effective in decreasing alcohol withdrawal symptoms, the number of bouts of withdrawal requiring standard medication treatment (lorazepam) and the amount of lorazepam required to control withdrawal bouts in individuals undergoing medical detoxification. Also, determine rates of subject recruitment and retention in the inpatient setting.

Participants: 80 alcohol dependent patients, 18-65 years of age, admitted for medical detoxification.

Procedures (methods): Subjects will be inpatients undergoing medical detoxification from alcohol. Oxytocin or placebo will be administered in a nasal spray twice daily in a randomized, double blind manner for three days. Withdrawal symptoms will be measured routinely at q4 hours and prn for length of hospital stay. Lorazepam will be given whenever withdrawal symptoms increase above specific parameters.

DETAILED DESCRIPTION:
Study Design: This will be a double-blind, placebo controlled comparison of the efficacy of twice daily intranasal administration of oxytocin and placebo (saline) in reducing alcohol withdrawal symptoms, the number of bouts of withdrawal during which symptoms are of sufficient magnitude requiring prn lorazepam treatment (see definitions below) and the amount of lorazepam required to resolve withdrawal bouts. Treatment group assignment will be random within each sex. Subjects will be patients admitted to (University of North Carolina (UNC) Hospitals or the Dix Clinical Research Unit (CRU) for medical detoxification. Each treatment group will be composed of up to 40 subjects. Dr. Hamer, the study statistician, will construct a randomization plan to randomize 80 subjects to 2 groups of 40 subjects each with a blocksize of 4. This will be a permuted blocksize as this is a blind study.

Procedures: Most patients who are admitted to the UNC Neuroscience Hospital Crisis Stabilization Unit, UNC Hospitals Family Practice or Hospitalist Services, or the Dix CRU for medical detoxification from alcohol will come in through the UNC Hospitals Emergency Department or Dorothea Dix Screening and Admissions during the late evening or early morning. Physical examination, medical and psychiatric history and lab tests (including complete blood count [CBC], magnesium, sodium, potassium, [blood urea nitrogen] BUN, creatinine, glucose, albumin, liver functions tests [ALT, AST, LDH, GGT], throid-stimulating hormone (TSH), B12, folate, urinalysis, urine toxicology screen and pregnancy test) are routinely obtained by the emergency department (ED)/ Dorothea Dix Screening and Admissions and/or inpatient unit during the admission process. Possibly in the UNC Hospitals ED/ Dorothea Dix Screening and Admissions and definitely after admission to these units, patients will have their vital signs (VSs) measured and their withdrawal symptoms quantified using the revised Clinical Institute Withdrawal Assessment for Alcohol scale (CIWA-Ar scale, Sullivan et al 1989) on the schedule in the standard alcohol detoxification order set in the UNC Hospital electronic medical records system (CPOE) system. The CRU at Dorothea Dix will use a hard copy version of the CIWA used in the CPOE at UNC Hospitals.

After consent is obtained, subjects will be randomly assigned to a treatment group (oxytocin or placebo). Prior to receiving their first intranasal treatment, an ECG will be obtained and blood drawn to obtain serum for assay of cytokine and allopregnanolone concentrations. Subjects also will rate their symptoms using the Alcohol Withdrawal Symptom Checklist (AWSC, Pittman et al 2007) prior to receiving their first test dose. These procedures will be done/overseen by research nurses or physicians. Subjects will usually receive their first intranasal test dose between 1000 and 1200 hours and will consist of 6 insufflations of Syntocinon Spray (approximately 24 IU) or placebo, with each insufflation given 30 seconds apart and alternating between nostrils. Test doses will be taken again at 1700 hr later that day (Admission Day 1) and at 0900 and 1700 hr on Admission Days 2 and 3. Oxytocin test treatments will be administered from 5 ml intranasal spray vials designed to deliver 0.1 ml metered volume per insufflation. The placebo treatments will be administered from 60 ml intranasal spray vials (each containing 30ml of solution) also designed to deliver 0.1ml metered volume per insufflation. Vials containing oxytocin and placebo spray will be blind labeled by the UNC Investigational Drug Service or the Dorothea Dix Hospital pharmacy. Research nurses or physicians will oversee subject self-administration of all intranasal test doses. After enrollment on admission day 1 and in the morning on admission days 2 and 3, subjects will be given multiple copies of the AWSC questionnaire and requested to complete one each time the unit nurses do CIWA ratings. These questionnaires will be retrieved by research staff the following morning. Shortly after the morning test dose on admission days 2 and 3, subjects will complete the Alcohol Craving Visual Analog Scales (ACVAS), the Penn Alcohol Craving Scale, and the Profile of Mood States (McNair et al, 1971). On these same admission days, research nurses will also draw (and subsequently process) blood serum samples to assay cytokine and allopregnanolone concentrations shortly after the morning test dose. Additional blood will be drawn after the morning test dose on admission day 2 to obtain serum for tests to be run in McLendon Laboratories (magnesium, chloride, calcium, sodium, potassium, BUN, creatinine, and liver function tests). Another electrocardiogram (ECG) will also be obtained shortly after the morning test treatment on admission day 2. Research staff will retrieve on a daily basis CIWA ratings and vital sign measurements obtained on each subject from their electronic medical record.

In all subjects, PRN lorazepam doses will be administered by mouth (PO) or intravenously (IV) (if subjects cannot take medication PO) whenever CIWA ratings are > 14 per the protocol in the standard alcohol detoxification order set in the UNC Hospital CPOE system. Lorazepam doses (1 - 4 mg) and frequency (q 2 -6 h) will be adjusted based on the severity of withdrawal symptoms. This same order set will be employed at the Dorothea Dix CRU.

ELIGIBILITY:
Inclusion Criteria:

* Daily consumption of 6 or more alcohol drinks/day for at least 2 weeks prior to admission.
* Only one of the following two conditions must be met:

  1. At least one prior episode 2 days or longer in duration which the subject experienced withdrawal symptoms that caused significant incapacitation.
  2. At least one prior inpatient or outpatient medical detoxification during which the subject exhibited withdrawal symptoms that sedative-hypnotic or anticonvulsant medication was required at least once on 2 consecutive days after cessation of or reduction in the use of alcohol following 2 weeks or more of heavily daily consumption (6 or more drinks/day).

Exclusion Criteria:

* Low literacy as indicated by an inability to read and understand the consent form.
* Dependence on substances other than alcohol, nicotine, caffeine or cannabis.
* History of alcohol withdrawal-related seizures, delirium tremens or hallucinations.
* Current or past alcohol-related medical complications (e.g. cirrhosis of the liver, esophageal varices, severe gastritis, hemoptysis, hematochezia or melena).
* Current delirium, disorientation to place or persons, seizures, acute or unstable psychosis or mania.
* Suicidal or homicidal ideation with strong intent, plans or recent attempt.
* Debilitating medical conditions (including AIDS, seizure disorder, emphysema, cancer and not well-controlled diabetes/hypertension) [HIV infection, diabetes, hypertension and asthma will not be grounds for exclusion]
* Diagnosis of amnesia, dementia, cognitive impairment or significant neurological symptoms.
* Low body weight (BMI<17).
* History of anorexia nervosa or bulimia in the past 2 years.
* Significant trauma, self injurious behavior or surgery in the previous 2 months
* Pregnancy; giving birth or breast-feeding in the past 6 months.
* Ingestion during the 2 weeks prior to this admission of much more alcohol/day than during previous drinking binges that preceded the onset of alcohol withdrawal symptoms.
* Ingestion of more than 450 ml of alcohol/day.
* Chronic treatment with benzodiazepines, barbiturates, anticonvulsants or stimulants
* Treatment/ingestion in the 72 hours prior to enrollment in the study with long half-life benzodiazepines or sedative hypnotic drugs.
* A blood alcohol level upon admission > 300 mg/dl.
* Well-documented history of inadequately treated baseline hypertension or tachycardia (SBP>150 or DBP>100 or P>110).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2010-07; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cort A Pedersen, M.D., Principal Investigator — The University of North Carolina, Chapel Hill, Department of Psychiatry
Locations (2):
- United States (2):
  - University of North Carolina Hospitals, Chapel Hill, North Carolina
  - Central Regional Hospital, Raleigh, North Carolina

REFERENCES:
- See also: UNC Department of Psychiatry — http://www.psychiatry.unc.edu/
- See also: UNC Department of Psychiatry Research — http://www.psychiatry.unc.edu/research

RESULTS

PARTICIPANT FLOW:
Groups:
- Intranasal Spray Without Oxytocin: Twice daily intranasal spray without oxytocin.
  intranasal spray without oxytocin: 6 insufflations (0.1 metered dose/insufflation) twice daily for 3 days
Period: Overall Study
Arm/Group | Intranasal Spray Without Oxytocin | Intranasal Oxytocin Spray
Started | 6 | 8
Completed | 4 | 7
Not Completed | 2 | 1
Not completed — Protocol Violation | 2 | 1

BASELINE CHARACTERISTICS:
Population: This was an intent to treat study in which data were collected and analyzed on all subjects in both treatment arms who were enrolled in the study and met eligibility criteria.
Groups:
- Total: Total of all reporting groups
Arm/Group | Intranasal Spray Without Oxytocin | Intranasal Oxytocin Spray | Total
Number analyzed (Participants) | 6 | 8 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.09 (8.32) | 42.23 (10.87) | 41.27 (14.67)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 8 | 14
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 5 | 7 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 5 | 8 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 8 | 14
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 8 | 14
CIWA-Ar score [Mean (Standard Deviation); unit: units on a scale] — Clinical Institute Withdrawal Assessment for Alcohol (CIWA) scale modified to include vital sign measurements. The CIWA scale measures each of 10 alcohol withdrawal symptoms between 0 and 6 (least to worst). Also in the modified CIWA score are ratings of body temperature (0-3, normal range to increasingly elevated), pulse (0-6), respirations (0-2), and diastolic blood pressure (0-6). So the range of possible total scores on the modified CIWA is 0-77.
  units on a scale | 9.25 (6.6) | 2.5 (1.4) | 4.5 (5.7)
Standard drinks/day over the past 2 weeks [Mean (Standard Deviation); unit: standard drinks/day] — A standard drink is defined as: 12-ounces of beer, 8-ounces of malt liquor, 5-ounces of wine, 1.5-ounces of 80-proof distilled spirits or liquor.
  standard drinks/day | 14.5 (1.7) | 17.7 (6.0) | 16.4 (4.7)

OUTCOME MEASURES:

1. Primary Outcome: Total Lorazepam Dosage (in Milligrams)
Description: Total lorazepam (in milligrams) required per subject to complete detoxification
Time Frame: Days 1 to 5
Measure: Mean (Standard Deviation); unit: milligrams of lorazepam
Arm/Group | Intranasal Spray Without Oxytocin | Intranasal Oxytocin Spray
Number analyzed (Participants) | 4 | 7
milligrams of lorazepam | 16.5 (4.4) | 3.4 (4.7)

2. Secondary Outcome: CIWA-Ar Scores
Description: Clinical Institute Withdrawal Assessment for Alcohol (CIWA) scale modified to include vital sign measurements. The CIWA scale measures each of 10 alcohol withdrawal symptoms between 0 and 6 (least to worst). Also in the modified CIWA score are ratings of body temperature (0-3, normal range to increasingly elevated), pulse (0-6), respirations (0-2), and diastolic blood pressure (0-6). So the range of possible total scores on the modified CIWA is 0-77.
Time Frame: days 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intranasal Spray Without Oxytocin | Intranasal Oxytocin Spray
Number analyzed (Participants) | 4 | 7
units on a scale | 11.8 (0.4) | 4.3 (2.3)

ADVERSE EVENTS:
Arm/Group | Intranasal Spray Without Oxytocin | Intranasal Oxytocin Spray
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/8
Other Adverse Events (participants affected / at risk) | 0/6 | 0/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intranasal Spray Without Oxytocin (N=6) | Intranasal Oxytocin Spray (N=8)
electrolyte abnormalities (Endocrine disorders) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No